CLINICAL TRIAL: NCT03192527
Title: A Phase I, Randomized, Placebo Controlled, Single Ascending Dose (SAD) Study of Recombinant Human Follicle Stimulating Hormone Fc Fusion Protein (KN015) in Healthy Female Volunteers
Brief Title: Single Dose Recombinant Human Follicle Stimulating Hormone Fc Husion Protein (KN015) in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alphamab Jilin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: KNJR-2017-001
Record Dates: First submitted 2017-06-14; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Infertility, Female
Keywords: KN015; Long-acting FSH
MeSH Terms: conditions — Infertility, Female | interventions — Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): KN015, Triptorelin
  Interventions: Drug: KN015; Drug: Triptorelin
- Arm B (Placebo Comparator): placebo, Triptorelin
  Interventions: Drug: Placebo; Drug: Triptorelin

INTERVENTIONS:
Drug: KN015 — experimental drug
  Arms: Arm A
Drug: Placebo — Comparator.
  Arms: Arm B
Drug: Triptorelin — The drug is used for down-regulation of endogenous FSH.

SUMMARY:
KN015,the active substance recombinant human Follicle Stimulating Hormone（FSH） Fc fusion protein, which belongs to the pharmaceutical class gonadotropins.KN015 is proposed for Assisted Reproductive Technology (ART) programs only. Its indication is Controlled Ovarian Stimulation （COS）in combination with a gonadotropin releasing hormone (GnRH) antagonist for the development of multiple follicles in women participating in an ART program. Due to its prolonged duration of FSH activity compared to conventional recombinant FSH (rFSH), a single subcutaneous injection of the recommended dose of KN015 may replace any daily rFSH preparation in a COS treatment cycle. This study is to evaluation of the safety, tolerability, pharmacokinetics and pharmacodynamics of KN015 in healthy Chinese female subjects.

DETAILED DESCRIPTION:
This is a phase I, randomized, placebo-controlled, single ascending dose, double blind parallel design, first-in-human study. The study design allows a gradual escalation of the dose-level with intensive safety monitoring to ensure the safety of the subjects. Dose escalation will continue until identification of MTD or up to a maximum dose of 100 μg. Tolerability, safety, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity characteristics of KN015 will be assessed in healthy female subjects. Eligible subjects will undergo down-regulation of endogenous FSH with a GnRH antagonist Triptorelin prior to receiving KN015.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent.
2. Agreed to take effective contraceptive measures during and 6 months after the end of the study period.
3. Age between 18 to 40 years (inclusive).
4. Body weight ≥45 kg, body mass index (BMI) of ≥18 and ≤28 kg/m2,
5. Regular menstruation cycle (25 to 34 days, inclusive).
6. Healthy female volunteer, normal findings in medical history and physical examinations.
7. Normal findings in sex hormone examinations unless the investigator considers an abnormality to be clinically irrelevant for this study.
8. Negative for human immunodeficiency virus (HIV) I and II tests, hepatitis B surface antigen (HBsAg), hepatitis C antibody and schaudinn's bacillus antibody at screening.
9. Normal uterus, presence of both ovaries, unless investigator considers an abnormality to be clinically irrelevant for this study.

Exclusion Criteria:

1. Historic abuse of alcoholic beverages and drugs. Smoke ≥5 cigarettes or the equivalent per day. Drug screen will include the minimum the following: amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, methadone, opiates.
2. History of hypersensitivity to FSH, or any documented or suspected allergy to KN015 or the excipients of the KN015 formulation, or hypersensitivity to luteinizing hormone releasing hormone agonist or something like that.
3. Any medical history of circulation, endocrine, nervous, digestive and respiratory systems, hematology, immunology, psychiatry and metabolic disorders and other serious disease history which can interfere with the test results of the study.
4. Polycystic ovary syndrome (PCOS).
5. Baseline of serum FSH ≥15 IU/L.
6. History of ovarian hyperstimulation syndrome (OHSS).
7. Experience in controlled ovarian stimulation (COS), or showed high response to FSH stimulation or the number of follicles over 11mm in diameter is more than 30.
8. The history of ovarian, breast, uterus, hypothalamus, and pituitary disease was determined by the investigators as clinical meaningful. Previous history of thrombosis or tending to suffer from thrombotic disease.
9. History of malignant disease.
10. Failing to comply with the special requirements of diet during study.
11. Participation in a clinical study within 3 months prior to the study.
12. Any medical condition that, in the opinion of the investigator, would interfere with safety of the subject or with the objectives of the study.
13. Abnormal physical examinational results which is determined as clinical significance by the researchers of the study.
14. Abnormal vital signs and clinical significance.
15. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >1.5 x ULN.
16. Thyroid dysfunction which clinical significance by researchers of the study.
17. Other abnormal laboratory tests with clinically relevance.
18. Abnormal electrocardiogram [ECG] findings.
19. III/IV class endometriosis, submucous myoma of uterus, endocrine abnormalities within 6 months prior to the study.
20. Abnormal imaging examination and clinical significance judged by researchers of the study.
21. Pregnancy or lactation period.
22. Alcohol and urine drug screening positive. -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment(SAEs) and AEs of special interest. | From screening to up to 36 days
Maximum observed serum concentration (Cmax) of KN015 in healthy Chinese female subjects | within 0.5 hour pre-dose, 2,5,8,12,24,30,36,40,48,54,60,72,96h,120,144,168,240,288,336,504,672 hours post-dose.
Time of Maximum observed serum concentration (Tmax) of KN015 in healthy Chinese female subjects. | within 0.5 hour pre-dose, 2,5,8,12,24,30,36,40,48,54,60,72,96h,120,144,168,240,288,336,504,672 hours post-dose.
Adjusted geometric means of area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUC(0-T)) for KN015. | within 0.5 hour pre-dose, 2,5,8,12,24,30,36,40,48,54,60,72,96h,120,144,168,240,288,336,504,672 hours post-dose.
Adjusted geometric means of area under the serum concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) for KN015. | within 0.5 hour pre-dose, 2,5,8,12,24,30,36,40,48,54,60,72,96h,120,144,168,240,288,336,504,672 hours post-dose.
Serum Half-life (T-HALF) of KN015 in healthy Chinese female subjects. | within 0.5 hour pre-dose, 2,5,8,12,24,30,36,40,48,54,60,72,96h,120,144,168,240,288,336,504,672 hours post-dose.
Serum clearance (CL) of KN015 in healthy Chinese female subjects. | within 0.5 hour pre-dose, 2,5,8,12,24,30,36,40,48,54,60,72,96h,120,144,168,240,288,336,504,672 hours post-dose.
Volume of distribution at steady state (VSS) of KN015 in healthy Chinese female subjects. | within 0.5 hour pre-dose, 2,5,8,12,24,30,36,40,48,54,60,72,96h,120,144,168,240,288,336,504,672 hours post-dose.

SECONDARY OUTCOMES:
The number of follicles after dosing. | screening,-1,2,4,6,8,11,15,22,29,36 days post-dose
The size of follicles after dosing. | screening,-1,2,4,6,8,11,15,22,29,36 days post-dose
Determination of serum concentrations of FSH, E2, LH and P after dosing. | From screening to up to 36 days
Percentage of participants with anti-KN015 antibody. | -1,8,15,36 days post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Chuangchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Fan Y, Gao L, Wang B, Xu T, Wu M, Liu J, Zhu X, Li X, Chen H, Li C, Wang M, Liu C, Mao Y, Yang M, Ding Y. The effect of a single escalating dose of long-acting recombinant human follicle-stimulating hormone Fc fusion protein (KN015) on healthy, pituitary-suppressed women: first-in-human and randomized study on its pharmacokinetics, pharmacodynamics, and tolerability. Expert Opin Investig Drugs. 2022 Nov;31(11):1255-1263. doi: 10.1080/13543784.2022.2151434. Epub 2022 Dec 20. PMID 36537742